CLINICAL TRIAL: NCT04336605
Title: Killing Pain - Use of Analgesic, Sedative and Anxiolytic Medication and the Development of Psychiatric Illness in Adolescents
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Oslo University Hospital (Other); The Change Factory (Unknown); Norwegian Council for Mental Health (Other); The Dam Foundation (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Synne O. B. Stensland, Principal Investigator (MD, PhD), Norwegian Center for Violence and Traumatic Stress Studies
Other Study IDs: Killing Pain; A pill for the pain (Other: NKVTS)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: PTSD; Psychiatric Illness; Prescription Drug Dependence; Addiction
Keywords: PTSD; Psychiatric Illness; Prescription drugs; Addiction; Adolescents
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Disorders; Behavior, Addictive | interventions — Aging; Growth and Development; Prescription Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young-HUNT: The young-HUNT study is a renowned, representative, population-based study where all adolescents living in the Nord-Trøndelag county have been invited to participate in four subsequent waves, from 1995 to 2019. Information about the study can be found here: https://www.ntnu.edu/hunt/young-hunt. In this study data from the Young-HUNT1-4 studies (1995-2019) will be linked to longitudinal, individual data from the Norwegian prescription Database (NorPD) (2004-2020), providing a unique, longitudinal dataset in which research questions will be explored. To obtain good, reliable follow-up data and outcome measures for the young-HUNT3 participants (2006-2008) the investigators will additionally include longitudinal data from the HUNT4 study of young adults (2017-2019); applicable for those participating in both the YoungHUNT3 and the YoungHUNT4.
  Interventions: Other: Age & Development; Other: Socioeconomy; Other: Traumatic Events; Other: Psychosocial conditions; Other: Lifestyle; Other: Chronic conditions; Other: Somatic symptoms; Other: Psychological symptoms; Other: Non-prescription analgesics; Other: Prescription drugs

INTERVENTIONS:
Other: Age & Development — Age, sex, pubertal onset and development
Other: Socioeconomy — Family structure and economy
Other: Traumatic Events — Violence and other traumatic events
Other: Psychosocial conditions — Family/social support
Other: Lifestyle — Physical activity, BMI, nutrition, smoking …
Other: Chronic conditions — I.e. Epilepsy or juvenile rheumatoid arthritis ...
Other: Somatic symptoms — Headache, pain, sleep disturbances ...
Other: Psychological symptoms — PTSS, anxiety, depressive symptoms & loneliness ...
Other: Non-prescription analgesics — Non-prescription analgesics
Other: Prescription drugs — Analgetic, sedative & anxiolytic medication

SUMMARY:
Prescription of analgesic, sedative, and anxiolytic medication for children and adolescents is increasing in Western countries. In recent decades, rates have also increased in Norway, despite a relatively restrictive prescription practice. Analgesics, sedatives, and anxiolytics are among the medications most commonly prescribed to young people by general practitioners and others. Overuse of such medication adversely impacts individual and societal health, social and economic measures. For example, the risk of chronification of pain, development of addiction, and dropout from school and the workforce is high. Epidemiological research has largely failed to integrate vulnerable, young service users' perspectives in planning, interpretation and dissemination of results. This has resulted in limited identification of potential causes for the increasing exposure to prescription and overuse of analgesics and other addictive drugs among of children and adolescents, and the long-term consequences this may have for morbidity and addiction in early adulthood. Knowledge of early risk factors and plausible causal mechanisms is crucial for the development of timely and effective interventions to prevent inappropriate prescriptions in clinical practice.

This prospective, longitudinal cohort study examines the use of analgesic, sedative, and anxiolytic medication among about 25,000 children throughout adolescence and young adulthood (1995 to 2020), specifically addressing changes in prescription over time, and early risk factors for the prescription of addictive drugs in adolescence and young adulthood and the subsequent development of mental health disorders.

DETAILED DESCRIPTION:
Linking data from the renowned, representative, population-based Nord-Trøndelag Health studies of adolescents (Young-HUNT, 1995-2019) to longitudinal, individual data from the Norwegian prescription Database (NorPD) (2004-2020) provides a unique, longitudinal dataset which will be examined in this study. Thus, the study design allows for examination of early predictors, risk factors, and potential causal mechanisms of prescription drug (analgesic, sedative, and anxiolytic medication) overuse, and development of severe mental illness in young people.

The Young-HUNT3 (2006-2008) study is among the world's first representative health surveys of youth encompassing questions about violence and other traumatic events, self-reported somatic and psychological health measures, a clinical examination, and consent to linkage to longitudinal health registries. The Young-HUNT4 (2017-2019) additionally includes validated actigraphy measures of activity and sleep. The full cohort of adolescents living in Nord-Trøndelag county were invited to participate in each of the study waves (HUNT1-4). Participation rates have been exceptionally high ranging from 78-90%. During school hours, the youth answered a number of health-related questions, including items on: physical violence, sexual abuse, bullying, and a range of other traumatic events (in the youngHUNT3 and 4); diagnosed chronic disease such as epilepsy, migraine, or juvenile rheumatoid arthritis; somatic and psychological symptoms, including recurrent headaches, abdominal pain, other musculoskeletal pain, autonomic somatic symptoms, sleep difficulties, post-traumatic stress reactions, psychological distress (anxiety/depression), and loneliness; use of non-prescription analgesics; pubertal onset and developmental stage; lifestyle, such as physical activity and nutrition; socio-economic and psychosocial factors. The study additionally comprised a validated headache interview, and clinical anthropometric measures. The HUNT4 included a week's measure of activity and sleep by the use of actigraphs. Information on age and gender was obtained from the Norwegian National Population Registry.

Each Young-HUNT participant's 11-digit social security number will be linked to individual data in the NorPD at the Norwegian Institute of Public Health. The NorPD registers all prescription drugs dispensed from pharmacies in Norway, and the database therefore contains a complete overview of all prescription drugs dispensed to individual patients outside hospitals, since 2004. Non-prescription drugs and medicines purchased abroad are not registered. Registered drugs are classified according to the International Anatomical Therapeutic Chemical Classification System (ATC). In this study, the investigators include information on the number of dispensed prescriptions of drugs classified within the following ATC codes: M01 (anti-inflammatory and anti-rheumatic agents), N01A (anesthetics, general), N02 (analgesics; opioids, other analgesics, and antipyretics and migraine agents), N05 (psycholeptics; antipsychotics, anxiolytics, hypnotics and anxiolytics), N06 (psychoanaleptics; antidepressants, ADHD and nootropics, and psycholeptics in combinations) and N07B (drugs for addiction disorders) from 2004 up to time of linkage (2019/2020).

To obtain good, reliable follow-up data and outcome measures for the young-HUNT3 participants (2006-2008) the investigators will additionally include longitudinal data from the HUNT4 study of young adults (2017-2019); applicable for those participating in both the YoungHUNT3 and the YoungHUNT4.

The data material provides a unique opportunity to study the following research questions:

1. Prevalence and comorbidity of migraine, other headache, chronic widespread pain, fatigue, insomnia and posttraumatic stress reactions and related risk profiles among adolescents.
2. How do discrepancies in risk & comorbidity profiles differentially affect young peoples' risk of analgesic, sedative, and anxiolytic medication overuse over time?
3. Do early somatic and psychological symptoms and self-medication in adolescence mediate risk of prescription drugs overuse in young people?
4. The role of early symptomatology and prescription drug overuse as predictive factors for development of severe psychiatric illness by young adulthood (age 29).

ELIGIBILITY:
Inclusion Criteria:

* All youth in Nord-Trøndelag county were invited to participate in four subsequent Young-HUNT study waves (1995-2019), https://www.ntnu.edu/hunt/young-hunt

Exclusion Criteria:

* None

Ages: 13 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All youth in Nord-Trøndelag county in Norway between 13-19 years were invited to participate in the four Young-HUNT study waves (1995-2019), and followed up after approximately 10 years between 2017-2020. In this study data from the Young-HUNT1-4 studies (1995-2019) will be linked to longitudinal, individual data from the Norwegian prescription Database (NorPD) (2004-2020), providing a unique, longitudinal dataset. To obtain good, reliable followup data for the young-HUNT3 participants (2006-2008) the investigators will additionally include longitudinal data of for those participating in both the YoungHUNT3 and the YoungHUNT4 (2017-2019).
Sampling Method: Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Prescription drugs | 2006-2020
  Analgetic, sedative & anxiolytic medication
Psychiatric Illness | 2006-2020
  Medically treated severe mental illness, i.e. depression, psychosis, dependency or addiction disorders

CONTACTS AND LOCATIONS:
Overall Officials: Synne O Stensland, MD PhD, Principal Investigator — Norwegian Centre for Violence and Traumatic Stress Studies
Locations (1):
- Norwegian Centre for Violence and Traumatic Stress Studies, Oslo, Norway

REFERENCES:
- [Derived] Baumann-Larsen M, Zwart JA, Dyb G, Wentzel-Larsen T, Stangeland H, Storheim K, Stensland SO. Killing pain? A prospective population-based study on trauma exposure in childhood as predictor for frequent use of over-the-counter analgesics in young adulthood. The HUNT study. Psychiatry Res. 2023 Sep;327:115400. doi: 10.1016/j.psychres.2023.115400. Epub 2023 Aug 1. PMID 37574601
- [Derived] Stangeland H, Handal M, Skurtveit SO, Aakvaag HF, Dyb G, Wentzel-Larsen T, Baumann-Larsen M, Zwart JA, Storheim K, Stensland SO. Killing pain?: a population-based registry study of the use of prescription analgesics, anxiolytics, and hypnotics among all children, adolescents and young adults in Norway from 2004 to 2019. Eur Child Adolesc Psychiatry. 2023 Nov;32(11):2259-2270. doi: 10.1007/s00787-022-02066-8. Epub 2022 Aug 27. PMID 36030342